CLINICAL TRIAL: NCT01688414
Title: Utility of Fluorescence and Photoacoustic Imaging Intraoperatively to Assist With Robotic Assisted Minimally Invasive Surgery
Brief Title: Imaging During Surgery in Diagnosing Patients With Prostate, Bladder, or Kidney Cancer
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI left Stanford
Sponsor: Stanford University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: VAR0083; NCI-2012-01654 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2012-09-12; First posted 2012-09-19 (Estimated); Last update posted 2014-07-29 (Estimated); Status verified 2014-07

CONDITIONS: Bladder Cancer; Kidney Tumor; Prostate Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms; Carcinoma, Renal Cell; Prostatic Neoplasms | interventions — Optical Imaging

ARMS (1):
- Diagnostic (fluorescence imaging, PAI) (Experimental): Patients undergo fluorescence imaging and PAI during robot assisted laparoscopic surgery.
  Interventions: Procedure: photoacoustic imaging; Procedure: fluorescence imaging; Procedure: robot-assisted laparoscopic surgery

INTERVENTIONS:
Procedure: photoacoustic imaging — Undergo PAI
  Other Names: optoacoustic imaging; PAI
Procedure: fluorescence imaging — Undergo fluorescence imaging
Procedure: robot-assisted laparoscopic surgery — Undergo robot-assisted laparoscopic surgery

SUMMARY:
This pilot clinical trial studies imaging during surgery in diagnosing patients with prostate, bladder, or kidney cancer. New diagnostic imaging procedures, may find prostate, bladder, or kidney cancer

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. The primary objective of this pilot study is to assess the ability of fluorescent imaging and photoacoustic imaging (PAI) in a clinical setting to distinguish benign from malignant tissue.

SECONDARY OBJECTIVES:

I. To qualitatively determine the possible benefit of PAI and fluorescent imaging over traditional white light imaging.

OUTLINE:

Patients undergo fluorescence imaging and PAI during robot assisted laparoscopic surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a pathologic confirmation of prostate cancer, bladder cancer, or kidney cancer based on previous biopsies or procedures OR a strong concern for a kidney malignancy based on computed tomography (CT) or magnetic resonance imaging (MRI) imaging
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients with a surgical history or anatomic variant that would preclude robot assisted laparoscopic approaches to their surgery (i.e. history of ventral hernia repair with mesh)
* Patients with medical co-morbidities who cannot tolerate laparoscopic surgery secondary to intra-abdominal carbon dioxide insufflation
* Patients with documented allergy or adverse drug reaction to indocyanine green or baseline serum creatinine greater than 1.5 mg/dL

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-09; Primary Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
Margin/lesion status determined by histopathology (cancer status [positive vs negative] as well as grade [Gleason grade 1-5 for prostate cancer, high vs low grade for bladder cancer, and Fuhrman grade 1-4 for kidney cancer]) | Up to 6 months after surgery
  The average lesion signal intensity on PAI and fluorescent imaging will be tested against the histology at pathological examination of the tissue sample.
Photoacoustic signal intensity (signal-to-noise ratio in the region of interest) | During the time of surgery
  The average lesion signal intensity on PAI and fluorescent imaging will be tested against the histology at pathological examination of the tissue sample. The distribution of signal intensity on PAI will be graphed as boxplot. The investigators will examine these parameters and compare them between malignant and benign cases using Wilcoxon rank-sum tests without making assumptions of normality.
Hemoglobin content (lesion total hemoglobin) as determined by photoacoustic measurements | During the time of surgery
  The distribution of signal intensity on hemoglobin content will be graphed as boxplots. The investigators will examine these parameters and compare them between malignant and benign cases using Wilcoxon rank-sum tests without making assumptions of normality.
Fluorescence intensity (signal-to-noise ratio in the region of interest) | During the time of surgery
  The distribution of signal intensity on fluorescence intensity will be graphed as boxplots. The investigators will examine these parameters and compare them between malignant and benign cases using Wilcoxon rank-sum tests without making assumptions of normality.
Oxygen saturation (percent oxygen saturation in region of interest) as determined by photoacoustic measurements | During the time of surgery
  The distribution of signal intensity on oxygen saturation will be graphed as boxplots. The investigators will examine these parameters and compare them between malignant and benign cases using Wilcoxon rank-sum tests without making assumptions of normality.

SECONDARY OUTCOMES:
Subjective operator determined characteristics for ease of identification of pedicle, NV bundle, and lymph nodes (prostate cancer patients) | During the time of surgery
  Descriptive statistics will be used to describe the operator determined secondary endpoints of the utility of each different imaging modality (i.e. white light, PAI, and fluorescence imaging).
Subjective operator determined characteristics for ease of identification of pedicle, ureter, and lymph nodes (bladder cancer patients) | During the time of surgery
  Descriptive statistics will be used to describe the operator determined secondary endpoints of the utility of each different imaging modality (i.e. white light, PAI, and fluorescence imaging).
Subjective operator determined characteristics for ease of identification of hilum and tumor (kidney cancer patients) | During the time of surgery
  Descriptive statistics will be used to describe the operator determined secondary endpoints of the utility of each different imaging modality (i.e. white light, PAI, and fluorescence imaging).

CONTACTS AND LOCATIONS:
Overall Officials: Mark Gonzalgo, Principal Investigator — Stanford University